CLINICAL TRIAL: NCT01189188
Title: Ultrasound Guidance for Radial Arterial Blood Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2010/RGG-03; 2010-A00714-35 (Other: ANSM)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Radial Artery; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With ultrasound guidance (Experimental): In this group of patients, ultrasound guidance will be used when drawing blood from the radial artery.
  Interventions: Procedure: Artery puncture with ultrasound guidance
- Without ultrasound guidance (Active Comparator): In this group of patients, no ultrasound guidance will be used when drawing blood from the radial artery.
  Interventions: Procedure: Artery puncture without ultrasound guidance

INTERVENTIONS:
Procedure: Artery puncture with ultrasound guidance — Ultrasound device will be used to locate artery for puncture.
  Arms: With ultrasound guidance
Procedure: Artery puncture without ultrasound guidance — Blood drawn from radial artery according to conventional procedure, without ultrasound guidance.
  Arms: Without ultrasound guidance

SUMMARY:
The investigators aim to determine if ultrasound guidance results in improved technique when drawing blood via a radial artery puncture.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed consent
* The subject is affiliated with a social security system
* Health status necessitates an arterial blood sample for diagnostic, prognostic or therapeutic reasons

Exclusion Criteria:

* The subject is participating in another study
* The subject is in a study exclusion period determined by a previous study
* The subject is under guardianship
* The subject refuses to sign consent
* Impossible to correctly inform the patient
* The patient is pregnant, breastfeeding, or parturient
* Allergies to one or more of the following: methyl, propylbenzoate, propylene glycol, chlorhexidine gluconate
* Contraindication for an arterial puncture (at the radial artery)
* Cardio-respiratory arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09-25 (Actual); Study Completion 2010-09-25 (Actual)

PRIMARY OUTCOMES:
Is only one puncture attempt necessary to attain the radial artery? yes/no | maximum two hours

SECONDARY OUTCOMES:
The number of puncture attempts required to attain the radial artery | maximum two hous
Visual Analog Scale score for pain felt by the patient (0.0 to 10.0) | Maximum two hours
Visual Analog Scale score for patient satisfaction (0.0 to 10.0) | Maximum two hours
Visual Analog Scale score for health professional satisfaction (0.0 to 10.) | Maximum two hours
Presence / absence of a hematoma at the site of puncture | two hours
Presence / absence of other complications | Two hours

CONTACTS AND LOCATIONS:
Overall Officials: Romain Genre-Grandpierre, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, France

REFERENCES:
- [Result] Bobbia X, Grandpierre RG, Claret PG, Moreau A, Pommet S, Bonnec JM, Bayard RP, Lefrant JY, Muller L, de La Coussaye JE. Ultrasound guidance for radial arterial puncture: a randomized controlled trial. Am J Emerg Med. 2013 May;31(5):810-5. doi: 10.1016/j.ajem.2013.01.029. Epub 2013 Mar 25. PMID 23535230
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140